CLINICAL TRIAL: NCT01906632
Title: Gene Expression Profiling of Malignant Tumor Predict the Therapeutic Response of DC-CIK Immunotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, Director, Capita Medical University Cancer Center, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMC
Record Dates: First submitted 2013-07-21; First posted 2013-07-24 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gene expression profile (Other)
  Interventions: Biological: DC-CIK Immunotherapy

INTERVENTIONS:
Biological: DC-CIK Immunotherapy

SUMMARY:
To investigate gene expression profile and immunological associated analysis relating to immunotherapy response of patients with malignant tumor after DC-CIK immunotherapy.

DETAILED DESCRIPTION:
1. The patients with malignant tumor are treated with dendritic cells (DC) plus cytokine induced killer cells (CIK) .
2. Venous blood (4 ml) is collected from each subject and placed into tubes containing Ethylene Diamine Tetraacetic Acid(EDTA) before and after each treatment. Lymphocytes are sorted by Fluorescence Activated Cell Sorting(FACS) and stored at -80°C until processing.
3. The T-Cell Receptor/B-Cell Receptor gene expression is detected by micro-array。
4. Estimate Immunotherapy response, time to disease progression, survival rates and clinical benefit response on patients. Response is assessed using Response Evaluation Criteria in Solid Tumor Group (RECIST) guidelines. Degree of response is used to divide the cancers into two groups: sensitive and non-sensitive to immunotherapy.
5. Compare the gene expression profile between different immunotherapy response groups to explore the mechanism that predict the DC-CIK immunotherapy response.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed with malignant tumor;
* Age: 18-80 years;
* an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* At least one measurable lesion according to the RECIST criteria;
* Adequate bone marrow, cardiac, liver, and renal function;
* Life expectancy ≥2 months;
* Not received other anti-tumor treatment
* Informed consent signed

Exclusion Criteria:

* previous history of other malignancies;
* Uncontrolled central nervous system metastases;
* Serious or uncontrolled concurrent medical illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
T-Cell Receptor/B-Cell Receptor gene expression | 3 month

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical Unvierstiy Cancer Center/ Beijing Shijitan Hospital, Beijing, China